CLINICAL TRIAL: NCT02016482
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Parallel-Arm, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Adalimumab for Treatment of Nail Psoriasis in Patients With Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Safety and Efficacy of Adalimumab in Subjects With Chronic Plaque Psoriasis and Nail Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-674; 2013-003275-36 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Nail Psoriasis; Plaque Psoriasis
Keywords: Nail Psoriasis; Plaque Psoriasis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (ADA) (Active Comparator): Period A: ADA 40 mg subcutaneous every other week (sc eow) for 25 weeks starting 1 week after initial loading dose of 80 mg. Period B: Placebo at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
  Interventions: Biological: Adalimumab; Other: Placebo
- Placebo (Placebo Comparator): Period A: Placebo sc eow for 25 weeks. Period B: ADA 80 mg sc at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
  Interventions: Biological: Adalimumab; Other: Placebo

INTERVENTIONS:
Biological: Adalimumab
  Other Names: ABT-D2E7; Humira
Other: Placebo

SUMMARY:
This study is being conducted to assess the safety and efficacy of adalimumab in participants with nail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have body surface area (BSA) ≥ 10% and a target fingernail Modified Nail Psoriasis Severity Index (mNAPSI) ≥ 8 at Week 0, OR BSA ≥ 5%, a target fingernail mNAPSI ≥ 8 and a total mNAPSI score of ≥ 20 at Week 0.
* Subject must have a Nail Psoriasis Physical Functioning Severity score of > 3, OR a Nail Psoriasis Pain Numeric Rating Scale (NRS) score of >3.
* Subjects must have a Physician's Global Assessment (PGA) of Fingernail Psoriasis and a PGA of Skin Psoriasis of at least moderate.
* Subject must have discontinued use of all systemic therapies for the treatment of psoriasis, or systemic therapies known to improve psoriasis for at least 4 weeks prior to Week 0, ustekinumab must have been discontinued at least 12 weeks prior to Week 0.
* Target fingernail must have mNAPSI score of ≥ 8.
* Adult subjects with clinical diagnosis of chronic plaque psoriasis (with disease duration of at least 6 months).

Exclusion Criteria:

* Prior adalimumab therapy.
* Diagnosis of other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of skin or fingernail psoriasis.
* Recent infection requiring treatment.
* Significant medical events or conditions that may put patients at risk for participation, including recent history of drug or alcohol abuse.
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study.
* History of cancer, except successfully treated skin cancer.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Williams, MD, Study Director — AbbVie

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Period A: Placebo subcutaneous every other week (sc eow) for 25 weeks. Period B: Adalimumab (ADA) 80 mg sc at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
- Adalimumab EOW: Period A: ADA 40 mg sc eow for 25 weeks starting 1 week after initial loading dose of 80 mg. Period B: Placebo at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
Period: Period A
Arm/Group | Placebo | Adalimumab EOW
Started | 108 | 109
Completed | 94 (56 participants early escaped to the end of Period A and 38 continued to the end of Period A.) | 94 (8 participants early escaped to the end of Period A and 86 continued to the end of Period A.)
Not Completed | 14 | 15
Not completed — Adverse Event | 3 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Lack of Efficacy | 2 | 1
Not completed — Other | 3 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Required Alternative/Prohibited Therapy | 0 | 1
Period: Period B
Arm/Group | Placebo | Adalimumab EOW
Started | 94 | 94
Completed | 81 | 87
Not Completed | 13 | 7
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lack of Efficacy | 6 | 4
Not completed — Other | 4 | 0
Not completed — Required Alternative/Prohibited Therapy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab EOW | Total
Number analyzed (Participants) | 108 | 109 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.16 (12.134) | 47.21 (11.858) | 46.69 (11.980)
Age, Customized [Number; unit: participants]
  < 40 years | 34 | 30 | 64
  40 to ≤ 64 years | 65 | 70 | 135
  ≥ 65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 87 | 96 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Total Fingernail Modified Nail Psoriasis Severity Index (mNAPSI) 75 Response at Week 26
Description: Each fingernail was assessed for psoriasis with mNAPSI, and the scores of all 10 fingernails were combined. Investigators assessed each nail abnormality for each of a participant's nails by grading 3 features or groups of features (pitting, onycholysis and oil-drop dyschromia, and crumbling) and noting the presence or absence of 4 features (leukonychia, splinter hemorrhages, hyperkeratosis, and red spots in the lunula). The range of possible scores was 0 to 130, with a score of 0 indicating absence of nail psoriasis and a score of 130 indicating the most severe nail psoriasis. A decrease in mNAPSI score indicates improvement. The mNAPSI 75 response is defined as at least 75% reduction from baseline in mNAPSI.
Time Frame: Week 26
Population: Intent-to-treat (ITT) Population in Period A: all participants who were randomized at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 3.4 | 46.6
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; For US regulatory purposes, ranked first secondary endpoint; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for strata. If zero frequency occurred, strata were dropped and p-value was calculated based on chi-square test (or adjusted chi-square test based on Campbell [2007]); Difference in percentage = 43.2, 95% CI 2-sided [32.8 to 53.6]

2. Primary Outcome: For United States (US) Regulatory Purposes: Percentage of Participants With a Physician's Global Assessment of Fingernails (PGA-F) of "Clear" or "Minimal" at Week 26
Description: The PGA-F is a 5-point scale used to assess fingernails separately for nail bed signs and nail matrix signs of disease. A global score of between 0 indicating clear, and 4 indicating severe, was separately assigned for nail bed involvement and nail matrix involvement. A participant's overall global score was the worse of the nail bed and nail matrix score. Data presents the percentage of participants with a PGA-F overall global score that met the definition of "clear" (0) or "minimal" (1) with at least a 2-grade improvement relative to Baseline at Week 26.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 6.9 | 48.9
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Ranked sixth secondary endpoint. For US regulatory purposes, this was the primary endpoint; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 42.0, 95% CI 2-sided [30.8 to 53.2]

3. Secondary Outcome: Percent Change From Baseline in Total Fingernail Nail Psoriasis Severity Index (NAPSI) Score at Week 26
Description: Each fingernail was assessed for nail matrix psoriasis and nail bed psoriasis with NAPSI and the scores of all 10 fingernails were combined. The range of possible scores was 0 to 80, with a score of 0 indicating absence of nail psoriasis and 80 indicating most severe nail psoriasis. A decrease in NAPSI score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | -11.5 (3.19) | -56.2 (3.12)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Ranked first secondary endpoint. For US regulatory purposes, ranked second secondary endpoint; Test type: Superiority or Other; p < 0.001, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean = -44.8, 95% CI 2-sided [-53.5 to -36.0]

4. Secondary Outcome: Percentage of Participants Achieving Total Fingernail mNAPSI Score of 0 at Week 26
Description: Each fingernail was assessed for psoriasis with mNAPSI, and the scores of all 10 fingernails were combined. The range of possible scores was 0 to 130, with a score of 0 indicating absence of nail psoriasis and a score of 130 indicating the most severe nail psoriasis. A decrease in mNAPSI score indicates improvement.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 0.0 | 6.6
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Ranked second secondary endpoint. For US regulatory purposes, ranked third secondary endpoint; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 6.6, 95% CI 2-sided [1.8 to 11.3]

5. Secondary Outcome: Percent Change From Baseline in Nail Psoriasis Pain Numeric Rating Scale (NRS) at Week 26
Description: An NRS was used to capture a participant's self-reporting of her/his worst fingernail pain and average fingernail pain due to fingernail psoriasis. The participant rated the severity of fingernail pain over the past 7 days on a scale from 0 indicating no pain, to 10 indicating severe pain. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | -1.1 (0.24) | -3.7 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Ranked third secondary endpoint. For US regulatory purposes, ranked fourth secondary endpoint; Test type: Superiority or Other; p < 0.001, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Percent Change = -2.6, 95% CI 2-sided [-3.3 to -2.0]

6. Secondary Outcome: Change From Baseline in Nail Psoriasis Physical Functioning Severity Score at Week 26
Description: Participants were asked to rate the impact of their fingernail psoriasis on their ability to perform physical tasks (eg, typing, housework, buttoning a shirt or blouse, picking up coins from a table, tying shoes, yard work, etc.) over the past 7 days on a scale of 0 indicating no impact on ability to perform physical tasks, to 10 indicating severe impact on ability to perform physical tasks. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -0.8 (0.24) | -3.7 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Ranked fourth secondary endpoint. For US regulatory purposes, ranked fifth secondary endpoint; Test type: Superiority or Other; p < 0.001, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = -2.9, 95% CI 2-sided [-3.6 to -2.2]

7. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in the Scalp Component of the Brigham Scalp Nail Inverse Palmo-Plantar Psoriasis Index (B-SNIPI) at Week 26
Description: The range of possible scores was 0 to 20 for scalp psoriasis, with a score of 0 indicating absence of psoriasis. A decrease in B-SNIPI score indicates improvement. Data presents the percentage of participants achieving 50% improvement in the scalp component of the B-SNIPI among participants with Baseline scalp score of ≥ 6.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Scalp psoriasis was assessed by B-SNIPI at Week 26 for participants enrolled under Protocol Amendment 1 in the US and Puerto Rico only. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 12 | 18
percentage of participants | 0.4 | 58.3
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Ranked fifth secondary endpoint. For US regulatory purposes, ranked sixth secondary endpoint; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 57.9, 95% CI 2-sided [33.8 to 82.0]

8. Secondary Outcome: Percentage of Participants Achieving "Clear" or "Minimal" in Nail Bed Component of the PGA-F at Week 26
Description: The PGA-F is a 5-point scale used to assess fingernails separately for nail bed signs and nail matrix signs of disease. A global score of between 0 indicating clear, and 4 indicating severe, was separately assigned for nail bed involvement and nail matrix involvement. A participant's overall global score was the worse of the nail bed and nail matrix score. Data presents the percentage of participants with a nail bed component of the PGA-F that met definition of "clear" (0) or "minimal" (1) among those with a Baseline nail bed component of "moderate" or "worse."
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had a Baseline nail bed component of "moderate" or "worse." Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 101 | 98
percentage of participants | 8.2 | 51.4
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 43.3, 95% CI 2-sided [31.3 to 55.2]

9. Secondary Outcome: Percentage of Participants Achieving "Clear" or "Minimal" in Nail Matrix Component of the PGA-F At Week 26
Description: The PGA-F is a 5-point scale used to assess fingernails separately for nail bed signs and nail matrix signs of disease. A global score of between 0 indicating clear, and 4 indicating severe, was separately assigned for nail bed involvement and nail matrix involvement. A participant's overall global score was the worse of the nail bed and nail matrix score. Data presents the percentage of participants with a nail matrix component of the PGA-F that met definition of "clear" (0) or "minimal" (1) among those with a Baseline nail matrix component of "moderate" or "worse."
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had a Baseline nail matrix component of "moderate" or "worse." Multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 99 | 102
percentage of participants | 8.5 | 53.3
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 44.8, 95% CI 2-sided [33.2 to 56.5]

10. Secondary Outcome: Percentage of Participants Achieving Target Fingernail mNAPSI Score of 0 at Week 26
Description: The target fingernail was assessed for psoriasis with mNAPSI. The range of possible scores was 0 to 13, with a score of 0 indicating absence of nail psoriasis and a score of 13 indicating the most severe nail psoriasis. A decrease in mNAPSI score indicates improvement.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 1.3 | 19.9
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 18.6, 95% CI 2-sided [10.6 to 26.6]

11. Secondary Outcome: Percentage of Participants Achieving Target Fingernail mNAPSI Score of ≤ 2 at Week 26
Description: as for outcome 10
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 7.3 | 43.3
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 36.0, 95% CI 2-sided [25.0 to 46.9]

12. Secondary Outcome: Percentage of Participants Achieving Total Fingernail mNAPSI Score of ≤ 2 at Week 26
Description: as for outcome 4
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 0.2 | 13.4
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 13.3, 95% CI 2-sided [6.5 to 20.0]

13. Secondary Outcome: Change From Baseline in Target Fingernail mNAPSI Score at Week 26
Description: as for outcome 10
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -2.1 (0.27) | -5.7 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — Across all strata, P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = -3.5, 95% CI 2-sided [-4.3 to -2.8]

14. Secondary Outcome: Percent Change From Baseline in Target Fingernail mNAPSI Score at Week 26
Description: as for outcome 10
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | -23.0 (2.92) | -61.9 (2.91)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -38.9, 95% CI 2-sided [-46.9 to -30.8]

15. Secondary Outcome: Change From Baseline in Total Fingernail mNAPSI Score at Week 26
Description: as for outcome 4
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -7.5 (1.78) | -36.1 (1.80)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -28.6, 95% CI 2-sided [-33.5 to -23.7]

16. Secondary Outcome: Percent Change From Baseline in Total Fingernail mNAPSI Score at Week 26
Description: as for outcome 4
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | -13.2 (3.06) | -63.3 (3.02)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -50.1, 95% CI 2-sided [-58.3 to -41.9]

17. Secondary Outcome: Percentage of Participants Achieving Total Fingernail NAPSI Score of 0 at Week 26
Description: as for outcome 3
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 0.0 | 7.5
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 7.4, 95% CI 2-sided [2.4 to 12.4]

18. Secondary Outcome: Percentage of Participants Achieving Target Fingernail NAPSI Score of 0 at Week 26
Description: The target fingernail was assessed for nail matrix psoriasis and nail bed psoriasis with NAPSI. The range of possible scores was 0 to 8, with a score of 0 indicating absence of nail psoriasis and 8 indicating most severe nail psoriasis. A decrease in NAPSI score indicates improvement.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 2.4 | 20.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 18.5, 95% CI 2-sided [10.1 to 26.8]

19. Secondary Outcome: Change From Baseline in Target Fingernail NAPSI Score at Week 26
Description: as for outcome 18
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -1.1 (0.21) | -3.6 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-3.1 to -1.9]

20. Secondary Outcome: Percent Change From Baseline in Target Fingernail NAPSI Score at Week 26
Description: as for outcome 18
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | -14.4 (3.50) | -54.6 (3.47)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -40.2, 95% CI 2-sided [-50.0 to -30.4]

21. Secondary Outcome: Change From Baseline in Total Fingernail NAPSI Score at Week 26
Description: as for outcome 3
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -6.7 (1.51) | -26.2 (1.47)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — Across all strata, P values were calculated from ANCOVA with stratum, Baseline value, and treatment in the model; LS Mean Difference = -19.5, 95% CI 2-sided [-23.6 to -15.3]

22. Secondary Outcome: Change From Baseline in Psoriasis Area Severity Index (PASI) Score at Week 26
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 to 72, with 0 indicating no psoriasis and 72 indicating very severe psoriasis. A decrease in PASI score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -0.9 (0.70) | -9.0 (0.70)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -8.1, 95% CI 2-sided [-10.0 to -6.1]

23. Secondary Outcome: Percent Change From Baseline in PASI Score at Week 26
Description: as for outcome 22
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | 2.4 (5.77) | -68.7 (5.70)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -71.2, 95% CI 2-sided [-87.3 to -55.0]

24. Secondary Outcome: Percentage of Participants Achieving PASI 75/50/90/100 Responses at Week 26
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 to 72, with 0 indicating no psoriasis and 72 indicating very severe psoriasis. PASI-75, 50, 90, and 100 responses are the percentage of participants with a Baseline PASI score ≥ 5 who achieved at least a 75%, 50%, 90%, or 100% reduction (improvement), respectively, from Baseline in PASI score at Week 26. A 100% reduction was considered complete clearance of psoriasis. Data presents the percentage of participants achieving PASI 75/50/90/100 responses at Week 26 among participants with a Baseline PASI score ≥ 5.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had a Baseline PASI score ≥ 5. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 95 | 97
percentage of participants
  PASI 75 | 13.8 | 64.8
  PASI 50 | 25.3 | 77.8
  PASI 90 | 7.1 | 48.0
  PASI 100 | 2.9 | 29.3
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; PASI 75; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 51.1, 95% CI 2-sided [38.6 to 63.5]
Statistical Analysis 2: Comparison: Placebo vs Adalimumab EOW; PASI 50; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 52.5, 95% CI 2-sided [39.9 to 65.0]
Statistical Analysis 3: Comparison: Placebo vs Adalimumab EOW; PASI 90; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 40.9, 95% CI 2-sided [29.0 to 52.9]
Statistical Analysis 4: Comparison: Placebo vs Adalimumab EOW; PASI 100; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 26.4, 95% CI 2-sided [15.8 to 36.9]

25. Secondary Outcome: Percentage of Participants Achieving Physician's Global Assessment of Skin Psoriasis (PGA-S) "Clear" or "Minimal" at Week 26
Description: The PGA-S is a 6-point scale used to measure the severity of skin disease at the time of the qualified investigator's evaluation of the participant. The degree of overall lesion severity was assessed, with 0 indicating cleared and 5 indicating severe. A decrease in PGA-S score indicates improvement. Data present the percentage of participants achieving a PGA-S of "clear" (0) or "minimal" (1) with at least a 2-grade improvement relative to Baseline at Week 26.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 11.2 | 63.4
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 52.2, 95% CI 2-sided [40.8 to 63.7]

26. Secondary Outcome: Percentage of Participants Achieving PGA-S of "Clear" at Week 26
Description: The PGA-S is a 6-point scale used to measure the severity of skin disease at the time of the qualified investigator's evaluation of the participant. The degree of overall lesion severity was assessed, with 0 indicating cleared and 5 indicating severe. A decrease in PGA-S score indicates improvement. Data present the percentage of participants achieving a PGA-S of "clear" (0) with at least a 2-grade improvement relative to Baseline at Week 26.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of participants | 4.0 | 28.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 24.8, 95% CI 2-sided [15.3 to 34.3]

27. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in the Inverse Psoriasis Component of the B-SNIPI at Week 26
Description: The range of possible B-SNIPI scores was 0 to 20 for inverse psoriasis, with a score of 0 indicating absence of psoriasis and a score of 20 indicating most severe psoriasis. A decrease in B-SNIPI score indicates improvement. Data presents the percentage of participants achieving 50% improvement in the inverse component of the B-SNIPI among participants with a Baseline inverse psoriasis score of ≥ 6.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had Baseline inverse psoriasis score ≥ 6. Inverse psoriasis was assessed for participants enrolled under Protocol Amendment 1 in the US and Puerto Rico only. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 11 | 12
percentage of participants | 0.5 | 90.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 90.4, 95% CI 2-sided [72.5 to 108.3]

28. Secondary Outcome: Change From Baseline in Total Body Surface Area (BSA) at Week 26
Description: BSA affected by psoriasis was measured by the physician selecting the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus 5 digits was to be assumed to be approximately equivalent to 1% BSA. Measurement of the total area of involvement by the physician was aided by imagining if scattered plaques were moved so that they were next to each other and then estimated the total area involved. A decrease in BSA affected by psoriasis indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percentage of affected BSA
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percentage of affected BSA | 0.4 (1.00) | -10.7 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -11.1, 95% CI 2-sided [-13.9 to -8.4]

29. Secondary Outcome: Percent Change From Baseline in Total BSA at Week 26
Description: as for outcome 28
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | 12.8 (6.08) | -67.8 (6.01)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -80.6, 95% CI 2-sided [-97.9 to -63.3]

30. Secondary Outcome: Percent Change From Baseline in Nail Psoriasis Pain NRS at Week 26
Description: as for outcome 5
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had an assessment (participants with an observed baseline value >0). Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 103 | 103
percent change | -18.0 (4.80) | -68.9 (4.70)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -50.9, 95% CI 2-sided [-64.0 to -37.8]

31. Secondary Outcome: Percent Change From Baseline in Nail Psoriasis Physical Functioning Severity Score at Week 26
Description: as for outcome 6
Time Frame: Baseline, Week 26
Population: as for outcome 30
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 105 | 104
percent change | -9.9 (5.51) | -67.6 (5.63)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -57.7, 95% CI 2-sided [-73.1 to -42.4]

32. Secondary Outcome: Change From Baseline in Nail Assessment in Psoriasis and Psoriatic Arthritis Quality of Life (NAPPA QoL) at Week 26
Description: Participants rated specific impacts of fingernail psoriasis on various aspects of their QoL over the past 7 days on a 5-point scale, with 0 indicating not at all, and 4 indicating very impactful. A participant's overall global score was the mean of all items and could range from 0 to 4, with 0 indicating no impact and 4 indicating most impact. A decrease in NAPPA QoL score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale | -0.4 (0.07) | -1.3 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.7]

33. Secondary Outcome: Percent Change From Baseline in Nail Assessment in NAPPA QoL at Week 26
Description: as for outcome 32
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
percent change | -11.7 (2.24) | -39.5 (2.23)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -27.7, 95% CI 2-sided [-33.9 to -21.6]

34. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 26
Description: Participants assessed symptoms and impacts of dermatologic diseases on their QoL over the past 7 days, with 0 indicating not at all, and 3 indicating very much. The range of possible DLQI scores was 0 to 30, with a score of 0 indicating no effect at all on a participant's life and a score of 30 indicating extremely large effect on participant's life. A decrease in DLQI score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had an assessment. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 93 | 94
units on a scale | -1.9 (0.60) | -8.0 (0.60)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -6.1, 95% CI 2-sided [-7.8 to -4.5]

35. Secondary Outcome: Percentage of Participants Achieving DLQI of 0 and 0/1 at Week 26
Description: Participants assessed symptoms and impacts of dermatologic diseases on their QoL over the past 7 days, with 0 indicating not at all, and 3 indicating very much. The range of possible DLQI scores was 0 to 30, with a score of 0 indicating no effect at all on a participant's life and a score of 30 indicating extremely large effect on participant's life. A decrease in DLQI score indicates improvement. Data presents the percentage of participants with a score of 0 (no effect) or 1 (little effect) at Week 26.
Time Frame: Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had an assessment. Multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 93 | 94
percentage of participants
  DLQI = 0 | 2.5 | 18.2
  DLQI = 0/1 | 3.7 | 30.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; DLQI = 0; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 15.7, 95% CI 2-sided [7.1 to 24.3]
Statistical Analysis 2: Comparison: Placebo vs Adalimumab EOW; DLQI = 0/1; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 27.1, 95% CI 2-sided [16.7 to 37.4]

36. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Nail Psoriasis (WPAI:NPSO) at Week 26
Description: The WPAI: NPSO assessed impact of fingernail psoriasis on work productivity and non-work activity limitation. Participants were asked during the past 7 days, how many hours did you miss from work because of problems associated with your fingernail psoriasis (absenteeism), during the past seven days, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study (presenteeism), how much did your fingernail psoriasis affect your productivity while you were working (overall work impairment), and much did your fingernail psoriasis affect your ability to do your regular daily activities, other than work at a job (activity impairment). Answers were rated on an 11-point scale, with 0 indicating "fingernail psoriasis had no effect on this" and 10 indicating "fingernail psoriasis completely prevented me from this." A decrease in the WPAI:NPSO score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline; n=number of participants with given assessment. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale
  Absenteeism; n=65, 74 | -1.0 (0.73) | -0.3 (0.65)
  Presenteeism; n=70, 77 | -3.4 (2.08) | -20.7 (2.06)
  Overall Work impairment; n=65, 74 | -6.2 (2.20) | -21.3 (2.05)
  Activity impairment; n=106, 108 | -1.8 (2.09) | -23.1 (2.18)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Absenteeism; Test type: Superiority or Other; p = 0.416, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [-1.0 to 2.5]
Statistical Analysis 2: Comparison: Placebo vs Adalimumab EOW; Presenteeism; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -17.3, 95% CI 2-sided [-22.9 to -11.6]
Statistical Analysis 3: Comparison: Placebo vs Adalimumab EOW; Overall work impairment; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -15.2, 95% CI 2-sided [-21.0 to -9.3]
Statistical Analysis 4: Comparison: Placebo vs Adalimumab EOW; Activity impairment; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -21.4, 95% CI 2-sided [-27.3 to -15.4]

37. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Health State Assessment at Week 26
Description: The EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the subject's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. A unique EQ-5D-5L health state is defined by combining the numeric level scores for each of the 5 dimensions and the total score is normalized from -0.594 to 1.000, with higher scores representing a better health state. An increase in the EQ-5D-5L total score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had an assessment. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 107 | 109
units on a scale | 0.0 (0.01) | 0.1 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = 0.1, 95% CI 2-sided [0.1 to 0.2]

38. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS) at Week 26
Description: The EQ-5D VAS records the participant's self-rated health status on a vertical graduated scale from 0 to 100, with 0 indicating the worst imaginable health state and 100 indicating the best imaginable health state. An increase in EQ-5D-5L VAS score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had an assessment. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 107 | 109
units on a scale | -0.1 (1.53) | 5.5 (1.53)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p = 0.012, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = 5.5, 95% CI 2-sided [1.2 to 9.8]

39. Secondary Outcome: Change From Baseline in Hospital Anxiety Depression Scale (HADS) at Week 26
Description: Participants rated their anxiety and depression over the past 7 days at Week 26. The range of possible scores was 0 to 21, with a score of 0 indicating absence of anxiety and depression and 21 indicating the most severe anxiety and depression. A decrease in HADS score indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline; n=number of participants with a given assessment. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 108 | 109
units on a scale
  HADS anxiety score; n=106, 109 | -0.1 (0.33) | -1.1 (0.33)
  HADS depression score; n=106, 108 | 0.0 (0.33) | -1.4 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; HADS anxiety score; Test type: Superiority or Other; p = 0.025, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = -1.1, 95% CI 2-sided [-2.0 to -0.1]
Statistical Analysis 2: Comparison: Placebo vs Adalimumab EOW; HADS depression score; Test type: Superiority or Other; p = 0.005, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = -1.3, 95% CI 2-sided [-2.3 to -0.4]

40. Secondary Outcome: Percentage of Participants With a New Diagnosis of Psoriatic Arthritis (PsA) During the Study
Description: The percentage of participants with a new diagnosis of PsA (ie, with an adverse event of PsA) during the study, among participants without PsA at Baseline.
Time Frame: up to Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and did not have PsA at Baseline. Observed cases.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 76 | 79
percentage of participants | 0 | 2
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p = 0.164, Chi-squared — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 2.5, 95% CI 2-sided [-0.9 to 6]

41. Secondary Outcome: Change From Baseline in Nail Psoriasis Quality of Life (Nail PsQoL) Score at Week 26
Description: Participants were asked how their fingernail psoriasis impacted their overall quality of life over the past 7 days on an 11-point scale, with 0 indicating no impact, and 10 indicating severe impact. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population in Period A: all participants who were randomized at Baseline and had an assessment. Multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab EOW
Number analyzed (Participants) | 107 | 109
units on a scale | -0.6 (0.23) | -3.3 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab EOW; Test type: Superiority or Other; p < 0.001, ANCOVA — P values were calculated from ANCOVA with treatment center stratum, Baseline value, and treatment in the model; LS Mean Difference = -2.8, 95% CI 2-sided [-3.4 to -2.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline through Week 52 +70 day follow up phone call; serious adverse events were collected from Screening through Week 52 + 70 day follow up call.
Groups:
- Placebo (Period A): Placebo sc eow for 25 weeks. Period B: ADA 80 mg sc at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
- Adalimumab EOW (Period A): ADA 40 mg sc eow for 25 weeks starting 1 week after initial loading dose of 80 mg.
- Placebo/Adalimumab EOW (Period B): Following Period A (placebo sc eow for 25 weeks), ADA 80 mg sc at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
- Adalimumab EOW/Adalimumab EOW (Period B): Following Period A (ADA 40 mg sc eow for 25 weeks starting 1 week after initial loading dose of 80 mg), placebo at Week 26 followed by ADA 40 mg sc eow from Week 27 through Week 51.
Arm/Group | Placebo (Period A) | Adalimumab EOW (Period A) | Placebo/Adalimumab EOW (Period B) | Adalimumab EOW/Adalimumab EOW (Period B)
Serious Adverse Events (participants affected / at risk) | 5/108 | 8/109 | 3/94 | 3/94
Other Adverse Events (participants affected / at risk) | 43/108 | 45/109 | 28/94 | 34/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period A) (N=108) | Adalimumab EOW (Period A) (N=109) | Placebo/Adalimumab EOW (Period B) (N=94) | Adalimumab EOW/Adalimumab EOW (Period B) (N=94)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1 | 1 | 0
ENDOCARDITIS (Infections and infestations) | 0 | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 2 | 0 | 0 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0 | 0 | 0
SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 1
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1 | 0 | 0
BLADDER SPHINCTER ATONY (Renal and urinary disorders) | 0 | 0 | 0 | 1
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period A) (N=108) | Adalimumab EOW (Period A) (N=109) | Placebo/Adalimumab EOW (Period B) (N=94) | Adalimumab EOW/Adalimumab EOW (Period B) (N=94)
DIARRHOEA (Gastrointestinal disorders) | 2 | 3 | 1 | 2
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 2 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 3 | 0 | 0
INJECTION SITE PAIN (General disorders) | 2 | 1 | 2 | 1
BRONCHITIS (Infections and infestations) | 0 | 2 | 3 | 2
GASTROENTERITIS (Infections and infestations) | 1 | 4 | 3 | 2
NASOPHARYNGITIS (Infections and infestations) | 10 | 6 | 9 | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 9 | 6 | 4
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 2 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 1 | 2
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 3 | 0 | 1 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 2
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
HEADACHE (Nervous system disorders) | 0 | 6 | 2 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1 | 0 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 6 | 1 | 4 | 1
HYPERTENSION (Vascular disorders) | 2 | 4 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to study design, a high percentage of participants randomized to the placebo arm early escaped from Period A and thus participated for a shorter duration than did participants in the active treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.